CLINICAL TRIAL: NCT01358747
Title: Randomized Phase III Study of a Treatment Driven by Early PET Response Compared to a Treatment Not Monitored by Early PET in Patients With Ann Arbor Stage III-IV or High Risk IIB Hodgkin Lymphoma
Brief Title: Study of a Treatment Driven by Early PET Response to a Treatment Not Monitored by Early PET in Patients With AA Stage 3-4 or 2B HL
Acronym: AHL 2011
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Collaborators: The Lymphoma Study Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel
Other Study IDs: Casasnovas PHRC N 2010
Record Dates: First submitted 2011-05-11; First posted 2011-05-24 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard arm (Active Comparator): Induction treatment: Patients will be treated by a BEACOPPesc regimen every 3 weeks for 4 cycles. A PET will be performed after 2 cycles of chemotherapy (PET2) with no decisional value, and after 4 cycles with decisional value. Consolidation treatment: depends on the reviewed PET4 result. In case of PET4 negative result, patient will received 2 additional cycles of BEACOPPesc, whatever the result of the PET2. In case of PET4 positive, the patient will be considered in treatment failure and proposed to a salvage therapy after pathologic confirmation of failure by biopsy of the hypermetabolic residual mass when possible.
  Interventions: Drug: BEACOPPesc
- Experimental arm (Experimental): Induction treatment: Patients will be treated by a BEACOPPesc regimen every 3 weeks for 2 cycles followed by a PET scan (PET2).
  After PET2 central review:
  * In case of positive PET2, the induction treatment will be completed by 2 additional cycles of BEACOPPesc
  * In case of negative PET2, the induction treatment will be completed by 2 cycles of ABVD delivered every 4 weeks. The first cycle of ABVD will start at day 21 of the second cycle of BEACOPPesc.
  Consolidation treatment: depends on the reviewed PET4 result In case of PET4 negative result, consolidation treatment will depends on PET2 results:
  * If PET2 was positive, patient will received 2 additional cycles of BEACOPPesc delivered every 3 weeks
  * If PET2 was negative, patient will received 2 additional cycles of ABVD delivered every 4 weeks In case of PET4 positive, the patient will be considered as treatment failure.
  Interventions: Drug: BEACOPPesc - ABVD - PET2

INTERVENTIONS:
Drug: BEACOPPesc
  Arms: Standard arm
Drug: BEACOPPesc - ABVD - PET2
  Arms: Experimental arm

SUMMARY:
All study treatments have proven efficacy in the treatment in Hodgkin lymphoma (HL). It is hoped that patients will achieve a good response to both induction therapies consisting either of 4 cycles of BEACOPPesc (Bleomycin, Etoposide, Doxorubicin, Cyclophosphamide, Vincristine, Procarbazine, and Prednisone) or 2 cycles of BEACOPPesc plus 2 cycles of ABVD (Adriamycine, Bléomycine, Vinblastine, Décarbazine).

The use of F-FDG Position Emission Tomography performed after 2 cycles of chemotherapy (PET2) in the experimental arm will help to stratify patients in order to restrict the BEACOPPesc therapy continuation to those patients who achieved only a partial response after 2 BEACOPPesc regimen and to allow a conventional dose ABVD chemotherapy strategy for PET2 negative patients. For all patients included in the trial the achievement of a good response to induction treatment will be checked after four cycles of induction treatment including a centrally reviewed PET assessment

Patients will be randomized after verification of eligibility and before the start of the protocol treatment.Patients will be randomly assigned to the standard treatment arm not monitored by early PET, or the experimental treatment arm driven by the PET2 result.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a first diagnosis of classical Hodgkin lymphoma according to world health organization (WHO) criteria excluding nodular lymphocyte predominant subtype
* Age of 16 to 60 years
* No previous treatment for Hodgkin lymphoma
* Ann Arbor stages:

IIB with mediastinum/thorax ≥0.33 or extra nodal localization III IV

* Baseline 18-FDG PET scan (PET0)(F-FDG Positon Emission Tomography) performed before any treatment with at least one hypermetabolic lesion
* Eastern Cooperative Oncology Group (ECOG) performance status < 3
* With a minimum life expectancy of 3 months
* Having previously signed a written informed consent
* The patient must be covered by a social security system (in France)

Exclusion Criteria:

* Pregnant or lactating women
* Men and women of childbearing potential not practicing an adequate method of contraception during the study treatment and at least 3 months after the last study drug administration
* Any history of cancer or cancer treatment during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma
* Uncontrolled infectious disease, including active HBV (hepatitis B virus) infection defined by either detection of HBs Antigen or presence of anti HBs antibody without detectable anti HBc antibody.
* HIV (Human immunodeficiency virus), HCV (hepatitis C virus) or HTLV (Human T-lymphotropic virus) serology positivity
* Abnormal liver (bilirubin > 2,5 N) function unless abnormalities are due to AHL 2011 Protocol Version n°1.2_ 09/02/11_approved on March 11, 2011 EudraCT n°2010-022844-19 4 / 73 Hodgkin lymphoma
* Abnormal renal (Creatinin > 150 μmol/L) function unless abnormalities are due to Hodgkin lymphoma
* Leukopenia < 2 G/l or thrombopenia <100 G/l unless abnormalities are due to Hodgkin lymphoma
* Severe cardio-pulmonary, or metabolic disease interfering with normal application of protocol treatment:
* Left Ejection Ventricular Fraction <50%
* Respiratory insufficiency prohibiting bleomycin use
* Uncontrolled diabetes mellitus leading to impossibility to perform PET scan
* Impossibility to perform a baseline PET (PET0) before randomization and treatment beginning
* Incapable person

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2011-05

PRIMARY OUTCOMES:
Progression free survival | 5 years
  Evaluate by PFS at 5 years the non-inferiority of a chemotherapy of a therapeutic strategy driven by PET with a ABVD conventional dose chemotherapy for patients reaching a negative PET after 2 cycles of BEACOPPesc, compared to a treatment not monitored by early PET delivering 6 cycles of BEACOPPesc.

CONTACTS AND LOCATIONS:
Overall Officials: René-Olivier CASASNOVAS, MD, Principal Investigator — CHU Dijon
Locations (96):
- Belgium (16):
  - ZNA Stuivenberg, Antwerp
  - Clinique sud Luxembourg, Arlon
  - RHMS, Baudour
  - Az Sint Jan, Bruges
  - Hôpital Erasme, Brussels
  - Ucl Bruxelles, Brussels
  - Grand hôpital de Charleroi, Charleroi
  - Hôpital Jolimont, Haine-Saint-Paul
  - AZ Groeninge, Kortrljk
  - chu Ambroise Paré, Mons
  - Clinique St Joseph, Mons
  - Clinique ST Pierre, Ottignies
  - AZ Delta, Roeselare
  - Centre Hospitalier Wallonie Picarde, Tournai
  - CH tourelle Peltzer, Verviers
  - Chu Mont Godinne, Yvoir
- France (80):
  - CHU Angers, Angers
  - CH Antibes, Antibes
  - CH Victor Dupouy, Argenteuil
  - CH d'Arras, Arras
  - CH Avignon - Hopital Duffaut, Avignon
  - Hopital de Bayonne, Bayonne
  - CHG Béziers, Béziers
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CH du Dr Duchenne, Boulogne-sur-Mer
  - CH de Bourg en Bresse, Bourg-en-Bresse
  - CH Jacques-Coeur, Bourges
  - Hôpital Morvan- CHU Brest, Brest
  - Ch Brive, Brive-la-Gaillarde
  - CHU de Caen-Côte de Nacre, Caen
  - Centre François Baclesse, Caen
  - Clinique du Parc, Castelnau-le-Lez
  - Hôpital de Chalon, Chalon-sur-Saône
  - CH Chambéry, Chambéry
  - Hopital Antoine Beclere, Clamart
  - Hôpital d'instruction des Armées Percy, Clamart
  - Hopitaux Civil de Colmar - Hopital Pasteur, Colmar
  - CH Sud Francilien, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - CHU Dijon - Hopital du Bocage, Dijon
  - CH de Dunkerque, Dunkirk
  - Chd Vendee, La Roche-sur-Yon
  - Hopital Saint Louis, La Rochelle
  - CH de Versaille - Hopital Mignot, Le Chesnay
  - CH Chartres - Hopital Louis Pasteur, Le Coudray
  - Hopital Bicetre, Le Kremelin Bicetre
  - Clinique Victor HUGO, Le Mans
  - CHU du Mans, Le Mans
  - CH Lens, Lens
  - Chru Lille, Lille
  - CHU de Limoge - Hopital Dupuytren, Limoges
  - Clinique de la Sauvegarde, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Calmettes, Marseille
  - Hopital de la conception, Marseille
  - CH Meaux, Meaux
  - CH Marc Jacquet, Melun
  - CHR Metz - Hopital Bon Secours, Metz
  - CHU Saint-Eloi, Montpellier
  - CRLC Val D'Aurelle, Montpellier
  - CH Mulhouse - Hopital Muller, Mulhouse
  - Centre Catherine de Sienne, Nantes
  - CHU Hotel Dieu, Nantes
  - Hopital Américain de Paris, Neuilly-sur-Seine
  - Centre Antoine lacassagne, Nice
  - CHU Nice - Hopital de l'Archet, Nice
  - CHU Caremeau, Nîmes
  - CHR de la Source, Orléans
  - Hopital Soint-Antoine, Paris
  - Hôpital ST Antoine, Paris
  - Institut Curie - Hopital Claudius Régaud, Paris
  - Hopital Saint-Louis, Paris
  - Hopital de la Pitié Salpétrière, Paris
  - Hopital Cochin, Paris
  - Hopital Necker, Paris
  - CH de Pau, Pau
  - Hôpital St Jean, Perpignan
  - CHU Haut Leveque - Centre François Magendie, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CH Dubos, Pontoise
  - CH de la région d'Annecy, Pringy
  - CHU Reims - Hopital Robert Debré, Reims
  - Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Clinique Mathilde, Rouen
  - CH Yves Le Foll, Saint-Brieuc
  - Institut Curie - Hopital Huguenin, Saint-Cloud
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - CHU de Strasbourg-Hopital de Hautepierre, Strasbourg
  - Hôpital Bretonneau, Tours
  - CH de Troyes, Troyes
  - CH Valence, Valence
  - CHU Brabois, Vandœuvre-lès-Nancy
  - CH de Bretagne Atlantique, Vannes
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Casasnovas RO, Bouabdallah R, Brice P, Lazarovici J, Ghesquieres H, Stamatoullas A, Dupuis J, Gac AC, Gastinne T, Joly B, Bouabdallah K, Nicolas-Virelizier E, Feugier P, Morschhauser F, Delarue R, Farhat H, Quittet P, Berriolo-Riedinger A, Tempescul A, Edeline V, Maisonneuve H, Fornecker LM, Lamy T, Delmer A, Dartigues P, Martin L, Andre M, Mounier N, Traverse-Glehen A, Meignan M. PET-adapted treatment for newly diagnosed advanced Hodgkin lymphoma (AHL2011): a randomised, multicentre, non-inferiority, phase 3 study. Lancet Oncol. 2019 Feb;20(2):202-215. doi: 10.1016/S1470-2045(18)30784-8. Epub 2019 Jan 15. PMID 30658935
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Casasnovas RO, Bouabdallah R, Brice P, Lazarovici J, Ghesquieres H, Stamatoullas A, Dupuis J, Gac AC, Gastinne T, Joly B, Bouabdallah K, Nicolas-Virelizier E, Feugier P, Morschhauser F, Sibon D, Bonnet C, Berriolo-Riedinger A, Edeline V, Parrens M, Damotte D, Coso D, Andre M, Meignan M, Rossi C. Positron Emission Tomography-Driven Strategy in Advanced Hodgkin Lymphoma: Prolonged Follow-Up of the AHL2011 Phase III Lymphoma Study Association Study. J Clin Oncol. 2022 Apr 1;40(10):1091-1101. doi: 10.1200/JCO.21.01777. Epub 2022 Jan 6. PMID 34990281
- [Derived] Demeestere I, Racape J, Dechene J, Dupuis J, Morschhauser F, De Wilde V, Lazarovici J, Ghesquieres H, Touati M, Sibon D, Alexis M, Gac AC, Moatti H, Virelizier E, Maisonneuve H, Pranger D, Houot R, Fornecker LM, Tempescul A, Andre M, Casasnovas RO. Gonadal Function Recovery in Patients With Advanced Hodgkin Lymphoma Treated With a PET-Adapted Regimen: Prospective Analysis of a Randomized Phase III Trial (AHL2011). J Clin Oncol. 2021 Oct 10;39(29):3251-3260. doi: 10.1200/JCO.21.00068. Epub 2021 Jun 22. PMID 34156881